CLINICAL TRIAL: NCT04629937
Title: Clinical Evaluation of a Multipurpose CZT Camera in Gated Tomographic Radionuclide Angiography: a Head to Head Comparison With a Cardiac Dedicated CZT Device
Brief Title: Evaluation of Whole-body CZT Camera in Gated Tomographic Radionuclide Angiography
Acronym: STARGAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO 2020-20
Record Dates: First submitted 2020-11-10; First posted 2020-11-16 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Cardiac Function
Keywords: SPECT; gated tomographic radionuclide angiography; Multipurpose CZT camera; left ventricle ejection fraction; Radionuclide angiography

STUDY DESIGN:
Intervention Model Description: All patients will undergo SPECT acquisitions with both multipurpose CZT camera and cardiac dedicated CZT camera.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPECT acquisitions (Experimental): All patients will undergo SPECT acquisitions with both multipurpose CZT camera and cardiac dedicated CZT camera.
  Interventions: Other: SPECT acquisitions

INTERVENTIONS:
Other: SPECT acquisitions — All patients will undergo SPECT acquisitions with both multipurpose CZT camera and cardiac dedicated CZT camera.

SUMMARY:
Tomographic radionuclide angiography (or blood pool) is a reproducible method to evaluate left ventricular ejection fraction that is needed during oncological treatments or to evaluate cardiopathies.

Cardiac-dedicated CZT systems allowed dose or time reduction. Multipurpose CZT cameras have not yet been evaluated in this indication. Moreover, the impact of attenuation correction is not known.

DETAILED DESCRIPTION:
Tomographic radionuclide angiography is a simple, rapid and reproducible method of cardiac function measurement, including left (LVEF) and right (RVEF) ventricular ejection fractions.

In addition to cardiological indications, this examination is often performed as part of cardiac toxicity screening during the various oncological treatments. This indication is all the more true since the arrival of CZT gamma cameras dedicated to cardiological studies has made it possible to reduce injected activities, as well as examination times.

The multipurpose CZT camera allows tomoscintigraphic acquisitions to be carried out using CZT technology as well. Unlike the CZT gamma cameras dedicated to cardiological studies, this system can be used for the exploration of different organs, and also allows the realization of CT slices for attenuation correction.

Patients included in this study will be double scanned both on a dedicated cardiac CZT camera and on multipurpose CZT camera, with CT. LVEF and RVEF will be then compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our Nuclear Medicine department for evaluation of cardiac function.

Exclusion Criteria:

* Patients treated with chemotherapy within 12 days.
* Under 18 years old patients.
* Pregnant women or at risk of pregnancy.
* Breast feeding.
* Painful patients.
* Patients under guardianship.
* Patients in whom a standard examination is not feasible (agitation).
* Patients who do not benefit from a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Assessment of left and right ventricular volumes and ejection fraction. | Day 0
  Automatic quantification of left and right ventricular volumes, left ventricle ejection fraction (LVEF) and right ventricle ejection fraction (RVEF) using BPGs software (Cedars-Sinai Medical Center, Los Angeles, USA).

SECONDARY OUTCOMES:
Assessment of left and ventricular volumes and ejection fraction with attenuation correction. | Day 0
  Assessment of an attenuation map from low dose CT data. Automatic quantification of left and right ventricular volumes, LVEF and RVEF using BPGs software (Cedars-Sinai Medical Center, Los Angeles, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique THIBAULT, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'Orleans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Carver JR, Shapiro CL, Ng A, Jacobs L, Schwartz C, Virgo KS, Hagerty KL, Somerfield MR, Vaughn DJ; ASCO Cancer Survivorship Expert Panel. American Society of Clinical Oncology clinical evidence review on the ongoing care of adult cancer survivors: cardiac and pulmonary late effects. J Clin Oncol. 2007 Sep 1;25(25):3991-4008. doi: 10.1200/JCO.2007.10.9777. Epub 2007 Jun 18. PMID 17577017
- [Background] Curigliano G, Cardinale D, Suter T, Plataniotis G, de Azambuja E, Sandri MT, Criscitiello C, Goldhirsch A, Cipolla C, Roila F; ESMO Guidelines Working Group. Cardiovascular toxicity induced by chemotherapy, targeted agents and radiotherapy: ESMO Clinical Practice Guidelines. Ann Oncol. 2012 Oct;23 Suppl 7:vii155-66. doi: 10.1093/annonc/mds293. PMID 22997448
- [Background] Garcia EV, Faber TL, Esteves FP. Cardiac dedicated ultrafast SPECT cameras: new designs and clinical implications. J Nucl Med. 2011 Feb;52(2):210-7. doi: 10.2967/jnumed.110.081323. Epub 2011 Jan 13. PMID 21233190
- [Background] Garcia EV. Are SPECT measurements of myocardial blood flow and flow reserve ready for clinical use? Eur J Nucl Med Mol Imaging. 2014 Dec;41(12):2291-3. doi: 10.1007/s00259-014-2924-2. No abstract available. PMID 25311927
- [Background] Slomka PJ, Berman DS, Germano G. New cardiac cameras: single-photon emission CT and PET. Semin Nucl Med. 2014 Jul;44(4):232-51. doi: 10.1053/j.semnuclmed.2014.04.003. PMID 24948149